CLINICAL TRIAL: NCT01866228
Title: Impact of Treatment Consultation Recordings on Cancer Patient Outcomes: A Prospective, Parallel, Randomized Controlled Trial
Brief Title: Clinical Trial of the Impact of Treatment Consultation Recordings on Cancer Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Tom Hack, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H2013:085; 126049 (Other Grant/Funding Number: Canadian Institutes of Health Research/126049)
Record Dates: First submitted 2013-04-16; First posted 2013-05-31 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Brain Tumor; Neuroendocrine Cancer
Keywords: Consultation Recording; Brain Tumor; Neuroendocrine Cancer; Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Neuroendocrine; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Consultation Recording (No Intervention): Participant does not receive consultation recording
- Consultation Recording (Experimental): Participant receives consultation recording
  Interventions: Other: Consultation Recording

INTERVENTIONS:
Other: Consultation Recording
  Arms: Consultation Recording

SUMMARY:
The time period from diagnosis through to the end of treatment is challenging for patients. Patients need information, assistance with decision making, and emotional and social support to help cope with their diagnosis and treatment. The first meeting with the cancer doctor is especially anxiety-provoking for patients who will learn, for the first time, their treatment options and likelihood of being cured. This anxiety causes many patients to have difficulty remembering the important pieces of information that their cancer doctor tells them during this consultation. The main goal of this study is to demonstrate the benefits of giving cancer patients an audio-recording of their first consultation with their cancer doctor. The investigators will include newly diagnosed patients from cancer centres in Winnipeg and Calgary. The types of cancer that will be included in this study are brain and neuroendocrine. Patients with these types of cancer are more likely to have confused thinking, and therefore may have the most to gain from receiving their consultation recordings. The study will include 244 patients, and those who sign consent forms to participate will be assigned by chance to either receive their treatment consultation recording or not. Patients will receive their recording immediately after their consultation, and will be able to listen to the recording at any time either alone, or with family and friends. To figure out whether the consultation recording provides patients with benefits, the investigators will administer some questionnaires to patients at 1 week after the consultation, and again at 3 and 6 months after the consultation. These questionnaires will assess the following patient outcomes: i) anxiety and depression, ii) perception of being informed about the disease and treatment, iii) satisfaction with cancer care, iv) satisfaction with the doctor, and v) the extent to which patients are satisfied with their degree of involvement in treatment decision making. The investigators hypothesize that patients who receive their consultation recording will experience more benefits than patients who do not receive their consultation recording.

ELIGIBILITY:
Inclusion Criteria:

* presenting with a primary diagnosis of non-recurrent or metastatic brain, or neuroendocrine cancer
* 18 years of age or older
* able to read and communicate using the English language
* access to a computer to enable consultation playback

Exclusion Criteria:

* deemed by a treating clinician (or primary nurse for the treating clinician) to have any severe psychiatric condition or cognitive dysfunction that precludes provision of free and informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-06; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Control Preferences Scale at 1-week post-consultation | 1-week post-consultation
  Subjective report of actual role played in decision making.
Change from Baseline in Control Preferences Scale at 3-months post-consultation | 3-months post-consultation
  Subjective report of actual role played in decision making.
Change from Baseline in Control Preferences Scale at 6-months post-consultation | 6-months post-consultation
  Subjective report of actual role played in decision making.
Change from Baseline in Patient Satisfaction with Cancer Care Scale at 1-week post-consultation | 1-week post-consultation
Change from Baseline in Patient Satisfaction with Cancer Care Scale at 3-months post-consultation | 3-months post-consultation
Change from Baseline in Patient Satisfaction with Cancer Care Scale at 6-months post-consultation | 6-months post-consultation
Change from Baseline in PrestMan Satisfaction with Doctor Scale at 1-week post-consultation | 1-week post-consultation
Change from Baseline in PrestMan Satisfaction with Doctor Scale at 3-months post-consultation | 3-months post-consultation
Change from Baseline in PrestMan Satisfaction with Doctor Scale at 6-months post-consultation | 6-months post-consultation
Change from Baseline in Hospital Anxiety and Depression Scale at 1-week post-consultation | 1-week post-consultation
Change from Baseline in Hospital Anxiety and Depression Scale at 3-months post-consultation | 3-months post-consultation
Change from Baseline in Hospital Anxiety and Depression Scale at 6-months post-consultation | 6-months post-consultation
Change from Baseline in Perception of Being Informed Scale at 1-week post-consultation | 1- week post-consultation
Change from Baseline in Perception of Being Informed Scale at 3-months post-consultation | 3-months post-consultation
Change from Baseline in Perception of Being Informed Scale at 6-months post-consultation | 6-months post-consultation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Hack, PhD, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hack TF, Ruether JD, Pitz M, Thiessen B, Degner LF, Chateau D. Impact of consultation recordings on patient-reported outcomes in patients with brain tumors: a parallel randomized controlled trial. Support Care Cancer. 2021 Oct;29(10):5681-5690. doi: 10.1007/s00520-021-06038-7. Epub 2021 Feb 17. PMID 33595717